CLINICAL TRIAL: NCT03359967
Title: Changes in Intrathoracic Impedance During Sacubitril/Valsartan Treatment: CHILISALT Study
Brief Title: Changes in Intrathoracic Impedance During Sacubitril/Valsartan Treatment
Acronym: CHILISALT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Izmir (Other)
Responsible Party: Principal Investigator, Ugur Onsel Turk, MD, Cardiologist, Assoc. Prof. MD. Cardiologist, FESC, EHRA Cardiac Device Specialist, Central Hospital, Izmir
Other Study IDs: CH1HF
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Heart Failure With Reduced Ejection Fraction
MeSH Terms: interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Entresto tablet — Changes in intrathoracic impedance and other related parameters between before- and after Sacubitril/Valsartan treatment collected via previously implanted device algoritm. (OptiVol Fluid Index)

SUMMARY:
The CHILISALT Study aimed to explore the effect of angiotensin-neprilysin inhibition on intrathoracic impedance and -derived fluid index in HFrEF patients who had a device for cardiac resynchronization therapy and/or an implantable cardioverter-deﬁbrillator (ICD; Medtronic Inc., Minneapolis, MN) allowing continuous measurement of intrathoracic impedance.

DETAILED DESCRIPTION:
Background Cardiac implantable electronic devices (CIEDs) that are improving clinical outcomes in selected heart failure with reduced ejection fraction (HFrEF) patients also collect valuable diagnostic information from continuous monitoring of several physiological variables such as intrathoracic electrical impedance. Intrathoracic electrical impedance monitoring has been used as a tool to evaluate pulmonary congestion. Intrathoracic impedance is inversely correlated to pulmonary volume expansion and has been linked to cardiac ﬁlling pressures. Decreasing in intrathoracic impedance and -derived fluid indices such as OptiVol Fluid Index, has been shown to predict heart failure hospitalizations and all-cause mortality in patients with HFrEF. Furthermore, studies also have shown the usefulness of monitoring impedance to initiate timely interventions preventing decompensation.

In patients with symptomatic HFrEF, the PARADIGM-HF trial demonstrated that sacubitril/valsartan significantly reduced the primary endpoint of cardiovascular mortality and heart failure hospitalization, compared with enalapril. The rate of all-cause mortality was also significantly reduced. Subsequently, Sacubitril/Valsartan is recommended by current guidelines as foundational therapy for many patients with symptomatic HFrEF.

However as a natriuretic agent, effects of Sacubitril/Valsartan treatment on intrathoracic impedance and fluid index remains unclear.

Objective The CHILISALT Study aimed to explore the effect of angiotensin-neprilysin inhibition on intrathoracic impedance and fluid index values in HFrEF patients who were implanted with a device for cardiac resynchronization therapy and/or an implantable cardioverter-deﬁbrillator (ICD; Medtronic Inc., Minneapolis, MN) allowing continuous measurement of intrathoracic impedance and OptiVol Fluid Index. Main outcome parameters are the change in intrathoracic impedanceand OptiVol Index values between baseline (before Sacubutril/Valsartan treatment) and, 14th and 28th days of Sacubutril/Valsartan treatment.

Material and Methods CHILISALT Study will designed as national, multicentre, non-interventional, observational, single arm cohort study. Study population will identified from dedicated CIED Clinics from participating centres. Patients will eligible if they had already taking Sacubitril/Valsartan for ≥2 weeks and had been implanted with CIED for ≥3 months. Additionally, eligible patients must have a CIED before Sacubitril/Valsartan prescription date. Due to descriptive (proof of mechanism) design of the CHILISALT Study a formal population volume calculation will not be made. However, after minimum 24 patients included an interim analysis will be done in terms of changes in impedance values and other related parameters between baseline and after Sacubitril/Valsartan treatment. An independent data monitoring committee will decide to enrol or to finalize the study according to main outcome variable distribution. Main outcome parameters are the change in intrathoracic impedance and OptiVol Fluid index values between baseline (before Sacubutril/Valsartan treatment) and, 14th and 28th days of Sacubutril/Valsartan treatment. As a tool to evaluate pulmonary fluid status, intrathoracic impedance measuring quantiﬁes impedance changes. CIEDs measured intrathoracic impedance (ohms) using the RV-coil to can vector. Impedance-derived fluid index will obtained using a cumulative sum mathematical model that calculates the differences between impedance measured in ohms (measured impedance) and a reference impedance. OptiVol Fluid index will be expressed in ohm-days. It was demonstrated that the index value exceeded 60 ohm-days, the crossing of this threshold value predicted both increased morbidity and mortality. Other possible confounders such as change in body weight (kilogram), current diuretic dose (miligram per day), requirement of intravenous diuretic therapy (yes/no), and the change from baseline to 28th day of the treatment in the clinical summary score on the Kansas City Cardiomyopathy Questionnaire (KCCQ; on a scale from 0 to 100, with higher scores indicating fewer symptoms and physical limitations associated with heart failure) is selected as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patients will eligible if they had already taking Sacubitril/Valsartan for ≥2 weeks and had been implanted with CIED for ≥3 months. Additionally, eligible patients must have a CIED before Sacubitril/Valsartan prescription date.

Exclusion Criteria:

* Patients younger than 18 years.
* Patients who not taking or taking <2 weeks Sacubitril Valsartan
* Patients who had a CIED which not using OptiVol algoritm for impedance measurement.
* Patients with structural pulmonary disease
* Patients with obstructive sleep apnea syndrome who using a continuous positive airway pressure device
* Patients with CIED pocket abcess

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Heart Failure with Reduced Ejection Fraction and had a CIED using OptiVol Fluid Index for intrathoracic impedance measurement.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2018-02-12 (Estimated); Primary Completion 2018-06-29 (Estimated); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in intrathoracic impedance values (ohms) between baseline and 14th and 28th days of Sacubutril/Valsartan treatment | Baseline (1st day), 14 th day and 28th day. (Screening=-10 to -1 day, Enrollment (Baseline Visit), Visit 1 (14+/-2 days), Visit 2 (28+/-4 days)
  Main outcome parameter is the change in intrathoracic impedance values (ohms) measuring with a CIED using its RV-coil to can vector between baseline (before Sacubutril/Valsartan treatment) and, 14th and 28th days of Sacubutril/Valsartan treatment. (Baseline value minus 14th day value) (Baseline Value minus 28 th day value) (Ohms) ( Decreasing in intrathoracic impedance has been shown to predict heart failure hospitalizations and all-cause mortality in patients with HFrEF.
Change in OptiVol Index Values (ohm-days) between baseline and 14th and 28th days of Sacubutril/Valsartan treatment. | Baseline, 14th and 28th days of Sacubitril/Valsartan treatment
  Change in Optivol Index values (ohm-days) measuring with a CIED using its RV-coil to can vector between baseline (before Sacubutril/Valsartan treatment) and, 14th and 28th days of Sacubutril/Valsartan treatment. (Baseline value minus 14th day value) (Baseline Value minus 28 th day value) (Ohm-days) Decreasing in intrathoracic impedance derived fluid indices such as OptiVol Fluid Index, has been shown to predict heart failure hospitalizations and all-cause mortality in patients with HFrEF.

SECONDARY OUTCOMES:
Change in body weight (kilogram) | Baseline, 14 th day and 28 th day
  Differences in Morning Body weight (kilogram) at fasting state between baseline and 14 th, 28 th days of Sacubitril/Valsartan treatment.
Change in cumulative diuretic dose (miligram per day) | Baseline, 14 th day, and 28 th day
  Changing of personal, current cumulative diuretic dose ( Between baseline and 14 th, 28 th days of Sacubitril/Valsartan treatment)
Requirement of intravenous diuretic therapy | Baseline, 14 th day, and 28 th day
  Requirement of intravenous a loop diuretic due to congestive status (inpatient and/or outpatient) (Admission times)
Change in the clinical summary score on the Kansas City Cardiomyopathy Questionnaire (KCCQ). | Baseline, 28 th day
  Change from baseline to 28th day of the treatment in the clinical summary score on the Kansas City Cardiomyopathy Questionnaire (KCCQ) (on a scale from 0 to 100, with higher scores indicating fewer symptoms and physical limitations associated with heart failure)

IPD SHARING:
Plan to Share IPD: No